CLINICAL TRIAL: NCT01238419
Title: Clinical Assessment of Physiotulle Dressing Compared to Urgotul Dressing in the Treatment of Leg Ulcer
Brief Title: Physiotulle vs Urgotul in the Treatment of Leg Ulcer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR010WS
Record Dates: First submitted 2010-10-27; First posted 2010-11-10 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2010-10

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotulle (Experimental)
  Interventions: Device: Physiotulle
- Urgotul (Placebo Comparator)
  Interventions: Device: URGOTUL

INTERVENTIONS:
Device: Physiotulle — Physiotulle is a non adherent dressing, composed of a polyester fabric impregnated with hydrocolloid particles (CMC) suspended in vaseline
  Arms: Physiotulle
Device: URGOTUL — Urgotul is an non occlusive dressing comprising of a polyester mesh impregnated with hydrocolloid particles dispersed on a petroleum jelly matrix
  Arms: Urgotul

SUMMARY:
The aim of this study is to assess the pain at removal of Physiotulle dressing in comparison with that of Urgotul dressing in patients presenting a venous (or predominantly) venous leg ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Patient of either sex over 18 who have not been declared legally incompetent and who having given his written informed consent
* Patient with venous or predominantly venous leg ulcer (ankle-brachial index > 0.8)
* Patient with venous or predominantly venous leg ulcer in granulation phase (granulation tissue > 70 %)
* Patient with venous or predominantly venous leg ulcer with low exsudate
* Patient with venous or predominantly venous leg ulcer with a wound surface between 4 cm² and 170 cm²
* Patient with venous or predominantly venous leg ulcer that has been treated with an appropriate compression in the two weeks prior to inclusion
* Patient available to be monitored for at least 4 weeks
* Patient able to answer questionnaires and particularly to evaluate his pain

Exclusion Criteria:

* Patient whose leg ulcer is locally infected (At least 3 of 5 clinical signs suggestive of infection *)* 5 signs suggestive of infection: pain, exsudate, smell, oedema, erythema
* Patient requiring an analgesic treatment for the care (before dressing removal)
* Patient whose ulcer belongs to angiodermatitis type or demonstrates a vasculitis
* Patient with arterial ulcer
* Patient with purely traumatic, infectious or neoplastic origin ulcer
* Patient with a diabetic neuropathy of lower limbs
* Patient with a known allergy to one of Physiotulle or Urgotul components
* Patient already participating in another clinical study
* Pregnant or breastfeeding patient

Patient who have been taking corticoids > 10mg / day or cytostatics by systematic way for the three months prior to inclusion

Patient who have undergone surgery of saphenous trunk in the two months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
pain at dressing removal | 4 weeks
  pain at dressing removal assessed by the patient immediately after dressing removal on a VAS scale

SECONDARY OUTCOMES:
Relative reduction of the area of the leg ulcer measured by planimetry at final point at week 4 compared to the area at inclusion | 4weeks
Number of patients with adverse events as a measure of safety and tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Locations (34):
- Denmark (3):
  - Bispebjerg ^Hospital, Bispebjerg, NV
  - Arhus Sygehus, Aarhus
  - Odense Universitets Hospital, Odense
- France (31):
  - Cabilet Medical, Abbeville
  - CHU Sud, Amiens
  - Cabinet Medical, Angoulême
  - Centre Hospitalier, Arras
  - Cabinet Médical, Bagnoles-de-l'Orne
  - CHU, Brest
  - CHU, Caen
  - Hôpital Manchester, Charlevilles Mézières
  - Centre Hospitalier de Douai, Douai
  - CHIVA, Foix
  - Hôpital de Freyming, Freyming Merleback
  - Centre Hospitalier, Haguenau
  - Hôpital Corention Celton, Issy-les-Moulineaux
  - CHD Les Oudairies, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - Cabinet Medical, Lille
  - Hôpital Dupuytren, Limoges
  - Cabinet Médical, Lunéville
  - Hôpital jacques Monod, Montivilliers
  - CHU Caremeau, Nîmes
  - Hôpital lariboisiere, Paris
  - CHRU La Miletrie, Poitiers
  - CH Cornouailles, Quimper
  - Clinique Mathilde, Rouen
  - Hôpital de Saint Gaudens, Saint-Gaudens
  - Centre hospitalier intercommunal, Saint-Germain-en-Laye
  - Cabinet Medical, Sarrebourg
  - HIA Sainte Anne, Toulon
  - Clinique Pasteur, Toulouse
  - CHRU Tours, Tours
  - CH, Valenciennes